CLINICAL TRIAL: NCT04681378
Title: A New Technique for Uterine Incision Closure at The Time of Cesarean Section: Does it Make a Difference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Nabih Elkhouly, associate professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID: 7-2016OBSGN17
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Cesarean Section; Wound Dehiscence
Keywords: Cesarean Section; Uterine Incision Closure

STUDY DESIGN:
Intervention Model Description: This trial enrolled 120 patients scheduled for primary cesarean delivery. Patients were randomized into either classical double layer uterine closure, purse string double layer uterine closure (Turan), or our new approach of uterine closure (double layer step up-step down technique). For short term comparison, transvaginal ultrasonography was planned for all patients 6 weeks after surgery
Who Masked: Participant, Outcomes Assessor
Masking Description: A computer-generated random numerical table (Randomization Generator Version 1.0) was used by our statistical department to prepare sealed opaque envelopes containing a group assignment. Three groups of envelopes-corresponding to the study groups were given to an anesthesia nurse. The nurse distributed envelopes to patients, alternating between groups during preanesthetic consultation. The patients were blinded the groups, and two authors performed the operations randomly. Another author who was blinded to the suturing technique performed all of the ultrasonographic examinations at 6 week follow up visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classical double layer closure (Active Comparator): a holding Vicryl 1-0 was placed in the in the left corner to stabilize and define the demarcation of the suture line. A continuous unlocked stitch beginning at the right corner was used, closing the whole thickness of the uterine wall, including the decidual layer. The second unlocked stitch was performed by Vicryl 1-0 in a lateral -lateral (horizontal) position, adapting the first layer. Up to three additional single sutures were added for hemostasis if required.
  Interventions: Procedure: double layer step up-step down technique
- Turan technique (Active Comparator): beginning in one corner, the incision is closed using Vicryl 1-0 stitch. The first layer is transversely passed through the inner myometrium-decidua line, and second layer is transversely passed through outer myometrium-visceral line continuously in the form of a purse string closure. With this technique, the original string is returned to the starting point and tied with a knot. Following the double layered purse-string closure, the aperture left in the middle of the uterine incision is closed with one separate figure of eight suture
  Interventions: Procedure: double layer step up-step down technique
- Double layer step up-step down technique (Active Comparator): the incision is closed using Vicryl 1-0 stitch starting from one corner. The first layer is transversely passed through the inner myometrium-decidua line, and second layer is transversely passed through outer myometrium-visceral line continuously by alternating continuous stitches through the upper (step up) and the lower (step down) uterine flaps. The original string is returned to the starting point and tied with knot as in Turan technique. Following the double layered step up-step down closure, additional single sutures were added for hemostasis if required
  Interventions: Procedure: double layer step up-step down technique

INTERVENTIONS:
Procedure: double layer step up-step down technique — the incision is closed using Vicryl 1-0 stitch starting from one corner. The first layer is transversely passed through the inner myometrium-decidua line, and second layer is transversely passed through outer myometrium-visceral line continuously by alternating continuous stitches through the upper (step up) and the lower (step down) uterine flaps. The original string is returned to the starting point and tied with knot as in Turan technique. Following the double layered step up-step down closure, additional single sutures were added for hemostasis if required

SUMMARY:
The purpose of this study was to compare the short term operative outcomes of three different surgical techniques for uterine incision closure during cesarean section (CS).

This trial enrolled 120 patients scheduled for primary cesarean delivery. Patients were randomized into either classical double layer uterine closure, purse string double layer uterine closure (Turan), or our new approach of uterine closure (double layer step up-step down technique). For short term comparison, transvaginal ultrasonography was planned for all patients 6 weeks after surgery. Compared to group II and Group III, residual myometrial thickness was significantly thinner in group I (P< 0.001). The number of patients with uterine niche was 10 (50% of all scar defects) in group I whereas it was 4 (20%) in group II and 6 (30%) in group III. Operative time was significantly longer in group II (P< 0.001). This led to our conclusion that Turan technique and our new approach are associated with thicker myometrial thickness and less frequency of uterine scar defect than classical double layer uterine incision closure; however, our approach takes less operative time.

DETAILED DESCRIPTION:
The investigators performed single site randomized clinical trial that was conducted at department of Obstetrics and Gynecology, Menoufia University Hospital, which is a large tertiary center in the Delta region in Egypt. The study population consisted of 120 eligible pregnant women with a singleton first-time cesarean delivery without preterm rupture of membranes, contractions or cervical dilatations that were recruited from the inward section one day before surgery from January 2017 to April 2019; only 114 cases remained for analysis. The study was approved by our hospital ethics committee and a written consent was obtained from each participant woman after full explanation of the study design. No important changes occurred to the trial design after it began, and the CONSORT guidelines was observed and completed.

Exclusion criteria were: pregnant women who refused to participate, women under age of 18 years, history of previous CS or any other uterine surgery ( Hystrotomy , myomectomy, perforation),placenta previa, abruptio placenta, fibroids located in the cervical or the cervico-corporal border, presence of maternal disease ( diabetes mellitus, anemia, connective tissue disorders, uterine malformations), reoperation following the CS, and presence of chorioamnionits. Secondary exclusion criteria were the need for more than three additional single sutures for hemostasis.

One author evaluated all obstetric patients who applied to the delivery room within the study period and selected eligible cases. After excluding patients who did not meet the inclusion criteria and patients who refused to participate, all remaining patients were equally randomized into either classical double layer uterine closure (group I), purse string double layer uterine closure (Turan technique, group II), or our technique of double layer step up- step down uterine closure (group III).

A computer-generated random numerical table (Randomization Generator Version 1.0) was used by our statistical department to prepare sealed opaque envelopes containing a group assignment. Three groups of envelopes-corresponding to the study groups were given to an anesthesia nurse. The nurse distributed envelopes to patients, alternating between groups during preanesthetic consultation. The patients were blinded the groups, and two authors performed the operations randomly. Another author who was blinded to the suturing technique performed all of the ultrasonographic examinations at 6 week follow up visit.

All cesarean deliveries were performed under spinal anesthesia. An abdominal opening was made through a slightly curved transverse incision that was placed 3-4 cm above the symphysis pubis (Pfannestiel incision). The subcutaneous tissue was left untouched apart from midline. The rectus sheath was separated along its fibers and the rectus muscles pulled apart. Stretching with index fingers opened the peritoneum and the uterus was opened by transverse lower segment incision (Kerr incision), then the hole was enlarged between the index finger of one hand and the thumb of the other hand.

Classical double layer closure of uterine incision was performed as follows: a holding Vicryl 1-0 was placed in the in the left corner to stabilize and define the demarcation of the suture line. A continuous unlocked stitch beginning at the right corner was used, closing the whole thickness of the uterine wall, including the decidual layer. The second unlocked stitch was performed by Vicryl 1-0 in a lateral -lateral (horizontal) position, adapting the first layer. Up to three additional single sutures were added for hemostasis if required. The Turan technique may be summarized as follows: beginning in one corner, the incision is closed using Vicryl 1-0 stitch. The first layer is transversely passed through the inner myometrium-decidua line, and second layer is transversely passed through outer myometrium-visceral line continuously in the form of a purse string closure. With this technique, the original string is returned to the starting point and tied with a knot. Following the double layered purse-string closure, the aperture left in the middle of the uterine incision is closed with one separate figure of eight suture (Figure 1A). Our new approach can also be summarized as follows: the incision is closed using Vicryl 1-0 stitch starting from one corner. The first layer is transversely passed through the inner myometrium-decidua line, and second layer is transversely passed through outer myometrium-visceral line continuously by alternating continuous stitches through the upper (step up) and the lower (step down) uterine flaps. The original string is returned to the starting point and tied with knot as in Turan technique. Following the double layered step up-step down closure, additional single sutures were added for hemostasis if required (Figure 1B). Included in the surgical technique was uterine exteriorization. The visceral and parietal layers were left open and the rectus muscle was not stitched. The rectus sheath was stitched with a continuous unlocked no 1 Vicryl and subdermal was closed in all patients.

All patients received prophylactic intravenous antibiotics (Cefazolin sodium vial. 1gm, i.v) preoperatively to reduce the rate of wound infection. In addition, uterotonics (5 IU units of oxytocin) were given intravenously as a bolus, before manual removal of the placenta to prevent postpartum hemorrhage. During the surgery, one author recorded operative time from skin incision to skin closure, blood loss, type of uterine closure technique used, and Kerr incision length before and after suturing and whether additional sutures for hemostasis were needed.

All patients were discharged within 3 days of the operation and a detailed transvaginal ultrasound examination was planned for all patients 6 weeks after surgery. Examinations were performed with C8-4V endocavitary transducer with frequency of 4-8 MHz (Philips, HD11 XE Ultrasound system, USA). The uterus was visualized in a sagittal plane with both the endometrium and the cervical canal visible, the scar area was magnified and the outcome measures were obtained from a frozen image. The scar was then visualized in a transverse plane by carefully rotating the probe at the level of the scar. Our main variable for scar evaluation was residual myometrial thickness (RMT). The cesarean scar site was identified as a small triangular anechoic defect in the anterior wall of the uterus (uterine niche). In these patients RMT was measured from the top of niche to serosal surface. In patients without a scar defect RMT was measured from the delineation of the endometrium to the serosal surface at the level of CS scar and total myometrial thickness was measured at the myometrium adjacent to CS scar in all patients (Figure 2). If a scar defect was identified, investigators measured in a sagittal plane its height (distance from the base/anterior lining of the endometrium to the apex) and width (W) at its base. The length of the defect at its base in a transverse axis (distance between the proximal and distal parts of the myometrium of the anterior uterine wall) was also recorded.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with a singleton prior cesarean section
* first-time cesarean delivery
* without preterm rupture of membranes, contractions or cervical dilatations

Exclusion Criteria:

* women under age of 18 years
* history of previous CS or any other uterine surgery
* placenta previa, abruptio placenta, fibroids located in the cervico-corporal border
* Maternal disease ( diabetes mellitus, anemia, connective tissue disorders, uterine malformations).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
residual myometrial thickness | 6 weeks after surgery
  The cesarean scar site was identified as a small triangular anechoic defect in the anterior wall of the uterus (uterine niche). In these patients RMT was measured from the top of niche to serosal surface. In patients without a scar defect RMT was measured from the delineation of the endometrium to the serosal surface at the level of CS scar and total myometrial thickness was measured at the myometrium adjacent to CS scar in all patients

REFERENCES:
- [Derived] Elkhouly NI, Abdelaal NK, Solyman AE, Elkelani OA, Elbasueny BF, Elhalaby AF. A new technique for uterine incision closure at the time of cesarean section: does it make a difference? J Obstet Gynaecol. 2022 Apr;42(3):416-423. doi: 10.1080/01443615.2021.1910636. Epub 2021 Jun 22. PMID 34155957